CLINICAL TRIAL: NCT04799821
Title: Eat Walnuts and Sleep Better: Exploring the Potential Role of Walnuts as Sleep-promoting Food and Their Impact on Body Composition
Brief Title: The Role of Walnut Consumption on Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: California Walnut Commission (Other)
Responsible Party: Principal Investigator, Dra. Maria Izquierdo-Pulido, Full Professor, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 600269
Record Dates: First submitted 2021-02-12; First posted 2021-03-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy Diet; Sleep
Keywords: Sleep quality; Walnuts; Body composition; Circadian rhythms
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Daily walnut consumption
  Interventions: Other: Walnut intake
- Control (Other): No walnut consumption
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — Participants will be asked to refrain from walnut intake and to follow an isocaloric meal plan that complies with the recommendations of a healthy Mediterranean-style eating pattern.
  Arms: Control
Other: Walnut intake — Participants will be asked to consume walnuts along with an isocaloric meal plan that complies with the recommendations of a healthy Mediterranean-style eating pattern.
  Arms: Intervention

SUMMARY:
Walnuts have a unique nutritional profile, including the sleep-regulating hormone melatonin, tryptophan, and omega-3 fatty acids, the two latest nutrients involved in melatonin and serotonin synthesis. Although it has been claimed that walnuts may improve sleep, to the investigators' knowledge, no studies have been conducted to objectively determine the impact of walnut consumption on sleep and overall well-being. Therefore, this study aims to investigate the effect of daily walnut consumption on sleep parameters (such as quality and duration). Secondarily, it aims to investigate the impact of daily walnut consumption on body composition, eating behavior, and well-being.

DETAILED DESCRIPTION:
The study to investigate the effect of daily walnut consumption on sleep quality will be conducted in an 18-week randomized crossover trial, in which participants will be initially assigned to intervention or control conditions for 8-weeks. After 2 weeks of washout, subjects will be crossed over to the alternate intervention and will continue for another 8 weeks. Note that throughout the whole study, each participant will attend 5 visits: 1 initial visit (baseline) and 2 visits in each one of the study conditions (intervention and control).

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-26 kg/m^2
* Habitual moderate exercise level
* No recent history of weight change exceeding 2.3kg (5lb) within the prior 3 months.

Exclusion Criteria:

* Nuts allergy
* Any acute or chronic diseases
* Smokers
* Any drugs or supplementations
* Any alimentary restrictions or specific diets
* Being a shift or night workers
* Being unable to give written informed consent.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in sleep onset latency from baseline to weeks 4, 8, 14, and 18 | Weeks 4, 8, 14 and 18
  Measured in hours of sleep with an actigraph (ActTrust, CONDOR, Brazil)
Changes in sleep efficiency from baseline to weeks 4, 8, 14, and 18 | Weeks 4, 8, 14 and 18
  Calculated in percentage as the ratio of total sleep time (TST) to time in bed (TIB).
  Sleep efficiency (percent) = (TST/TIB)*100
Changes in wake after sleep onset (WASO) from baseline to weeks 4, 8, 14, and 18 | Week 4, 8, 14, and 18
  Measured in minutes of WASO with an actigraph (ActTrust, CONDOR, Brazil)
Changes in sleep duration from baseline to weeks 4, 8, 14, and 18 | Weeks 4, 8, 14, and 18
  Measured in hours of sleep time with an actigraph (ActTrust, CONDOR, Brazil)
Changes in urinary 6-sulphaoxymelatonin from baseline to week 4, 8, 14 and 18 | Week 4, 8, 14 and 18
  Quantified using urine Melatonin-Sulfate ELISA kit

SECONDARY OUTCOMES:
Changes in body mass index (BMI) from baseline to weeks 4, 8, 14, and 18 | Weeks 4, 8, 14 and 18
  Calculated as weight (kg) divided by height (in squared meters), BMI= kg/m^2
Changes in body fat from baseline to weeks 4, 8, 14, and 18 | Weeks 4, 8, 14 and 18
  Measured as the percentage of body fat with a body composition analyzer (Inbody 120, Korea)
Changes in weight circumference from baseline to weeks 4, 8, 14, and 18 | Weeks 4, 8, 14 and 18
  Measured midway between the lower rib margin and the iliac crest with the subject standing and wearing only underwear, at the end of gentle expiration with an anthropometric tape (CESCORF, Brazil)
Changes in eating behavior from baseline to weeks 8 and 18 | Weeks 8 and 18
  To evaluate changes in eating behavior, the Spanish version of the Food Cravings Questionnaire will be used (Cepeda-Benito et al, 2000).
  This questionnaire evaluates 10 dimensions of eating behavior:
  * Having Intentions and Plans to Consume Food
  * Anticipation of Positive Reinforcement that may Result from Eating
  * Anticipation of Relief from Negative States and Feelings as a Result of Eating
  * Lack of Control over Eating
  * Thoughts or Preoccupation with Food
  * Having Intentions and Plans to Consume Food
  * Craving as a Physiological State
  * Emotions that may be Experienced Before or During Food Cravings or Eating
  * Cues that may Trigger Food Cravings
  * Guilt from Cravings and/or for Giving in to Them
  For each subscale, scores range from 0 to 5, with higher scores indicating a stronger sensation of craving.
Changes in well-being from baseline to weeks 8 and 18 | Weeks 8 and 18
  Well-being will be measured with the Spanish version of the WHO-5 Well-being Index (Lucas-Carrasco et. al. 2012).
  Scores range from 0 to 100, with higher scores indicating higher well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Izquierdo-Pulido, PhD, Principal Investigator — University of Barcelona
Locations (1):
- Torribera Campus, University of Barcelona, Santa Coloma de Gramenet, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.